CLINICAL TRIAL: NCT02753790
Title: Single Center, Phase II Study of Whole Brain Radiation Using IMRT to Spare the Hippocampus While Delivering Differential Doses to Subclinical Sites Versus Gross Disease for Treatment of Patients With Brain Metastases
Brief Title: Whole Brain Radiation Using IMRT for Patients With Brain Metastases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New Mexico Cancer Research Alliance (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INST 1409
Record Dates: First submitted 2016-04-20; First posted 2016-04-28 (Estimated); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Neoplasm Metastasis; Central Nervous System Metastases
Keywords: Brain; Metastasis; IMRT; Radiation; Cancer; Hippocampus; Intensity modulated radiotherapy; Quality of life; QOL
MeSH Terms: conditions — Neoplasm Metastasis; Neoplasms | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intensity Modulated Radiotherapy (IMRT) (Experimental): Radiation therapy to a dose of 60 Gray (Gy)/45 Gy to gross disease and 30 Gy to subclinical sites, delivered over 15 fractions
  Interventions: Radiation: Intensity Modulated Radiotherapy

INTERVENTIONS:
Radiation: Intensity Modulated Radiotherapy — Whole brain radiation using IMRT: 60 Gy to gross disease (planning treatment volume [PTV] 60) or 45 Gy to gross disease (PTV 45) and 30 Gy to subclinical sites (PTV 30) over 15 fractions.
  Patients will be treated Monday through Friday (5 days per week) for 3 weeks. Patients with either a single metastasis greater than 15 cubic centimeters (cm) or total volume of metastases greater than 26 cubic cm will receive the lower dose of 45 Gy to visible brain metastases. 45 Gy may also be prescribed per physician discretion.
  Gross disease which has received prior radiosurgery will receive 30 Gy.
  Other Names: IMRT

SUMMARY:
Some cancers can spread, or metastasize, to the brain. When they do, treatment often involves surgery and/or radiation. Optimal treatment of brain metastases would maximize disease control and minimize toxicity (or side effects), and improve the quality of life of patients. A common type of radiation used for brain metastases is called whole brain radiation, which treats not just the cancer that can be seen on scans (i.e., gross disease), but the smaller sites of cancer that may not be visible (i.e. subclinical disease). Fractionation is used to describe repetitive treatments in which small doses (fractions) of a total planned dose are given at separate clinic visits. The most common dosing regimen is 30 Gray (Gy), using 3 Gy per fraction over 10 fractions. Previous studies have suggested that using intensity modulated radiation therapy (IMRT) may be a safer way to deliver higher doses to gross disease and lower doses to the rest of the brain that may contain subclinical disease. This approach may spare the rest of the brain from radiation complications and side effects.

The goal of this study is to determine whether using IMRT to treat brain metastases is more effective than current standard whole brain radiation in controlling gross disease and whether patient quality of life and hair loss is improved compared to previous studies using whole brain radiation.

DETAILED DESCRIPTION:
This phase II clinical trial will utilize intensity modulated whole brain radiation therapy in order to deliver a smaller, yet effective dose for subclinical disease while giving a higher dose to gross disease for patients with more than one brain metastasis. In this study, a dose of 30 Gray (Gy) will be prescribed to subclinical sites and 60 or 45 Gy to visible brain metastases.

There is evidence from previous studies (including Radiation Therapy Oncology Group (RTOG) 0933) that hippocampal avoidance during whole brain radiotherapy using IMRT may decrease toxicity in the form of memory loss. Patients who had brain metastases within the region of hippocampal avoidance were not eligible for enrollment on RTOG 0933. In contrast, this study will include this group of patients since IMRT will be used to not only deliver higher doses to visible brain metastases even though they are located within the hippocampal avoidance region, but also to avoid the hippocampus itself. This approach may help to preserve memory function. Additionally, while temporary (and sometimes permanent) alopecia results from conventional whole brain radiation, IMRT spares the skin and possibly decreases the rate of hair loss. Dose to the scalp will be limited to as low as possible in order to decrease the risk of permanent alopecia in this study.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven diagnosis of a non-hematopoietic malignancy other than small cell lung cancer and germ cell malignancy within 5 years of registration. Patients with metastasis of unknown primary tumor are permitted.
* History/physical examination within 30 days prior to registration.
* Age ≥ 18 years
* Karnofsky performance status ≥ 70
* Ability to understand and the willingness to sign a written informed consent document.
* Women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Women of childbearing potential must have a negative qualitative serum pregnancy test ≤ 2 weeks prior to study entry. A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria: 1) Has not undergone a hysterectomy or bilateral oophorectomy; or 2) Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).
* More than one brain metastasis (qualifying measurable brain lesions are any contrast enhancing metastases identifiable by the physician).
* Patients who have undergone a resection for brain metastases will be eligible for participation if they have any residual metastases present on post operative MRI of the brain.

Exclusion Criteria:

* Patients with leptomeningeal metastases
* Plan for chemotherapy or targeted therapies during whole brain radiation or within 1 week of completing radiation therapy
* Contraindication to Magnetic Resonance (MR) imaging
* Serum creatinine > 1.4 mg/dl ≤ 30 days prior to study entry
* Prior radiation therapy to the brain besides radiosurgery
* Severe active comorbidities which would make the patient an unacceptable candidate for this clinical trial per physician discretion
* Patients with brain metastases involving the brainstem or chiasm
* Non English speaking patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-03-09 (Actual); Primary Completion 2021-04-22 (Actual); Study Completion 2022-04-10 (Actual)

PRIMARY OUTCOMES:
Overall response rate (ORR) | 3 months post-treatment
  Overall response rate (ORR) is the sum of the percentage of patients who achieve a complete response (CR) or partial response (PR). CR is defined as a total radiographic disappearance of all lesions with stabilization of the neurological examination after glucocorticoids have been stopped. PR is defined as a greater than 50% decrease in volume of all lesions as measured radiographically with improvement or stabilization of the neurological examination with stable glucocorticoid dose.

SECONDARY OUTCOMES:
Change in memory | 4 months post-treatment
  To assess change in memory, the Hopkins Verbal Learning Test-Revised (HVLT-R) will be administered prior to initiation of radiation (baseline) and at four months post-treatment. The test involves memorizing a list of 12 targets and recalling the 12 targets after a 20-minute delay (delayed recall or HVLT-R DR). Each patient will be his/her own control and the mean change in scores between baseline and four months will be calculated by subtracting the score at four months from the score at baseline and then dividing by the baseline score. A positive change indicates a decline in function. The mean change in scores will be reported.
Rate of permanent alopecia | 12 months post-treatment
  Alopecia (hair loss) will be assessed per National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE), version 4.03. Permanent alopecia is defined as CTCAE grade 2 (moderate; >50% normal for an individual that is readily apparent to others; a wig or hair piece is necessary if the patient desires to completely camouflage the hair loss; associated with psychosocial impact). The percentage of patients experiencing permanent alopecia will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Ben Liem, MD, Principal Investigator — University of New Mexico Comprehensive Cancer Center
Locations (1):
- Universtiy of New Mexico Comprehensive Cancer Center, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of New Mexico Comprehensive Cancer Center — http://www.cancer.unm.edu
- See also: New Mexico Cancer Care Alliance — http://www.nmcca.org